CLINICAL TRIAL: NCT04924634
Title: Stress Levels and Mental Well-Being Among Slovak Students During e-Learning in The COVID-19 Pandemic
Brief Title: Stress Levels and Mental Well-Being Among Slovak Students During e-Learning
Status: Completed | Type: Observational
Sponsor: The Opole University of Technology (Other)
Responsible Party: Sponsor
Other Study IDs: COVID_Slovak
Record Dates: First submitted 2021-06-08; First posted 2021-06-14 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: Anxiety State; Depression
Keywords: depression; e-Learning; COVID-19; anxiety
MeSH Terms: conditions — Anxiety Disorders; Depression; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Students: Students from 4 universities, regardless of field of study and academic year
  Interventions: Diagnostic Test: Stress Levels and Mental Well-Being assessment

INTERVENTIONS:
Diagnostic Test: Stress Levels and Mental Well-Being assessment — At the beginning of the summer semester of the 2020/2021 academic year, stress levels as well as symptoms of anxiety and depression were assessed in students at four universities.

SUMMARY:
Introducing restrictions on human contact has been effective in preventing the uncontrolled spread of COVID-19, however, it appears to have negatively impacted mental health. Psychological problems in different age groups occur with different intensity and duration of the pandemic. This study was aimed to assess the impact of introducing distance learning (e-Learning) on the stress levels and mental well-being among Slovak Students.

DETAILED DESCRIPTION:
Socially isolated young people, condemned to constant contact with the Internet, find themselves in sorrowful situations where their basic need were impossible. Previous studies report that university students report high levels of stress, anxiety, and depression, which affects student motivation and attitudes toward learning; however, to date, no such studies have been conducted on a population of Slovakian Students. This study considered 4 Slovak universities. Using standardized questionnaires, students' mental status during e-Learning was assessed at the beginning of the summer semester (February, March 2021).

ELIGIBILITY:
Inclusion Criteria:

* Students attending the course cycle

Exclusion Criteria:

* Inability to self-complete the research questionnaires;
* Psychiatric or psychological treatment, likewise taking medications that affect the psyche during the research project;

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Students participating in active learning
Sampling Method: Probability Sample
Enrollment: 3051 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-04-23 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale (PSS-10) | 20 minutes
  The PSS-10 is widely used for measuring psychological distress. It contains 10 questions on a five-point scale from 0 to 4. The higher the score, the greater the feeling of stress.
BDI | 20 minutes
  The BDI-II is a tool used to determine the degree of intensity of depressive symp-toms. The 21-item questionnaire consists of two parts: emotional and somatic. Depending on the number of points obtained, the severity of depression can be assessed. A range of 0-10 points indicates no depression, 11-27 indicates moderate mood disorder, and 28 indicates major depressive disorder. The cutoff for dividing patients into depressive and non-depressive subgroups was a score of 10, following the guidelines given by Beck et al.
Authors survey | 10 minutes
  The survey contains five sections on the impact of e-learning on various aspects of life. The survey responses were structured on a 5-point Likert scale from 1 to 5, where 1 refers to "strongly disagree" statement and 5 to "definitely agree". Questions were grouped into areas: Social life (3 questions), Education skills (4 questions), Eco-nomic field (2 questions), Nutrition habits and drugs (2 questions). The questionnaire showed satisfactory reliability with a Cronbach alpha of 0.82.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Education and Physiotherapy, Opole University of Technology, Opole, Poland

IPD SHARING:
Plan to Share IPD: No